CLINICAL TRIAL: NCT05552131
Title: A Prospective, Multicenter, Single-group, Target-value Clinical Trial to Evaluate the Safety and Efficacy of Coronary Lithotripsy Catheter System for Lumen Preconditioning in Moderate-to-severe Coronary Artery Calcification
Brief Title: Clinical Trial of T-wave™ Coronary Lithotripsy Catheter System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Zhonghui Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-T-01
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Moderate to Severe Calcified Coronary Artery Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary lithotripsy catheter system + drug-eluting stent (Experimental)
  Interventions: Device: T-wave coronary lithotripsy catheter system

INTERVENTIONS:
Device: T-wave coronary lithotripsy catheter system — Subjects who plan to receive possible interventional therapy meet all admission criteria and do not meet any exclusion criteria, and enter the screening stage of this clinical trial after signing informed consent. All subjects who sign the informed consent will be provided with a unique subject screening number. All subjects who met the inclusion criteria and did not meet the exclusion criteria were enrolled and lumen pretreated with a coronary shock catheter system followed by the implantation of drug-eluting stents.

SUMMARY:
A prospective, multi-center, single-group target value method was used in this study. According to the inclusion criteria stipulated in this trial protocol, > 3 medical device clinical trial institutions with the record of the State Food and Drug Administration were selected as clinical centers, and 190 cases were selected (the first case of each center was taken as the imported case. Follow-up was carried out according to the program process, but the results were analyzed separately. Moderate-to-severe calcified stenosis patients who met all the inclusion criteria and did not meet any exclusion criteria were enrolled into the study. Lumen pretreatment was performed using the coronary shock catheter system and drug-eluting stents were implanted.

Subjects were followed up immediately after surgery, before discharge, 30±3 days after surgery, and 6 months ±14 days after surgery to evaluate the safety and effectiveness of coronary lithotripsy catheter system for preconditioning patients with moderate and severe coronary artery calcification stenosis.

In this study, the success rate of postoperative surgery was used as the primary endpoint, and major cardiovascular and cerebrovascular adverse events within 30 days after surgery were used as the secondary endpoint.

After the completion of the primary endpoint evaluation of the project, it shall be submitted together with other data to the competent department of medical device approval for initial registration. At the same time, continue to complete the follow-up of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Subjects had primary coronary artery disease suitable for percutaneous coronary intervention (including stable or unstable angina pectoris and asymptomatic myocardial ischemia)
3. marker of myocardial injury： 3.1 For patients with unstable ischemic heart disease, the biomarker (CK-MB) must be within the normal range within 12 hours before surgery； 3.2 In patients with stable ischemic heart disease, biomarkers can be tested before or during surgery, and (CK-MB) must be within the normal range within 12 hours before or during surgery；
4. Patients were able to understand the content of the trial, volunteered to sign the informed consent, were willing to comply with the trial protocol, and had the ability to visit and check regularly;

Image inclusion criteria:

1. No stent has been implanted in the target lesion within 1 year, and no drug-eluting stent has been implanted within 5mm of the target lesion;
2. Single new stenosis of the left main artery of the target vessel, or of the anterior descending branch, right crown or circumflex branch (or its branches), with the following characteristics:

   1. Visual stenosis ≥70% and <100%; or
   2. Visual stenosis ≥50% but <70%, combined with evidence of clinical ischemia, such as typical clinical symptoms or positive tablet test results, or fractional flow reserve FFR≤0.80, or instantaneous waveform free ratio instantaneous wave-free ratio<0.90;
3. Moderate to severe calcification in the target lesion site is defined as:

   1. Angiography: Calcification can be detected in at least one location on either side of the arterial wall when the heart is beating or not under fluoroscopy before contrast medium injection; or
   2. Calcification ≥180° was present in at least one section by intravascular ultrasound.
4. The reference diameter of target vessels was between 2.5mm and 4.0mm;
5. Length of target lesion ≥5mm but ≤40mm;
6. Target vessels must have thrombolysis in myocardial infarction grade 3 before registration (can be evaluated after pre-dilation)
7. 0.014 inch guide wire can pass through the lesion;

Exclusion Criteria:

Basic condition (Cardiac function)

1. Left ventricular ejection fraction (LVEF) <40%;
2. New York Classification of Cardiac Function (NYHA) Class IV; Anatomical structure
3. There is a second lesion with an interval of more than 10mm and a stenosis degree of ≥50% in the same target vessel;
4. Target vessels were too circuitous, defined as the presence of two or more bends >90º or three or more bends >75º;
5. Definite or probable thrombus in the target vessel;
6. Evidence of aneurysm in the target vessel within 10mm of the target lesion;
7. The target lesion is located in the primary vessel that can only be reached by saphenous vein or arterial graft bypass;
8. There were restriction-limiting dissection with NHLBI (National Heart, Lung, and Blood Institute)grade ≥D in the target vessels before registration.
9. Chronic occlusive disease (CTO) : CTO exists in other main vessels outside the target vessel (anterior descending branch, circumflex branch, right crown) or CTO exists in any location of the target vessel.
10. Target lesions need to be pretreated with special balloons such as rotary grinding and spinous process balloon; Laboratory tests
11. uncontrolled severe hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure > 120 mmHg);
12. Acute myocardial infarction (MI) within the past 1 month, and/or signs of active myocardial ischemia at enrollment, including elevated troponin-I or T (with elevated CK), ischemic ECG changes, or chest pain;
13. Severe impairment of liver and kidney function, aminotransferase more than 3 times the upper limit of normal, creatinine > 2.5 mg/dL (221 μmol/L) or chronic renal failure requiring long-term dialysis; Note: In subjects with proven or suspected acute MI (as determined by the primary and secondary investigators), markers of myocardial injury must be evaluated prior to enrollment.

    Medical history and Others
14. 14. History of stroke or transient ischemic attack (TIA) within 30 days;
15. Patients with active peptic ulcer or upper gastrointestinal bleeding within 30 days;
16. Had undergone percutaneous coronary intervention within 14 days;
17. Patients who were scheduled to undergo a cardiovascular intervention within 30 days after this procedure;
18. Patients refuse or are not candidates for emergency coronary artery bypass grafting (CABG) surgery;
19. Drug-eluting stents have been implanted in target vessels within the past year;
20. Patients with known allergies or contraindications to the raw materials or drugs of the test products (such as antiplatelet drugs, anticoagulants, contrast agents);
21. Participating in other clinical trials;
22. The patient's expected survival was less than 1 year;
23. Women planning to have children during pregnancy, breastfeeding or clinical trials;
24. Factors that other researchers believe cannot be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of operation | Immediately after the procedure
  After the successful passage of the experimental medical device, the residual stenosis rate of the target lesion immediately after the implantation of the drug-eluting stent was less than 50% and no MACE(Major Adverse Cardiovascular Events) occurred in the hospital after the use of the coronary shock catheter system for lumen preparation.

SECONDARY OUTCOMES:
Success rate of contrast | Immediately after using the test control advice in treatment
  After successful passage of the experimental medical instruments, residual stenosis of the target lesion was < 50% after preconditioning and there were no serious angiographic complications, including flow limiting dissection (NHLBI grade D-F type)(NHLBI:National Heart, Lung, and Blood Institute) perforation, acute lumen occlusion, and persistent slow flow or no reflow.
Operation success rate 2 | Immediately after using the test control advice in treatment
  After lumen preparation using experimental medical instruments, residual stenosis rate of target lesion after drug eluting stent implantation was less than 50%, blood flow grading was TIMI level 3, and no MACE event occurred during hospitalization.
Residual stenosis rate of target lesions after pretreatment with experimental medical instruments | Immediately after the procedure
Residual stenosis rate of target lesions immediately after operation | Immediately after the procedure
Thrombolysis In Myocardial Infarction blood flow grading of target lesions immediately after operation | Immediately after the procedure
Major adverse cardiovascular events (MACE) event rate | Immediately after the procedure、30days、180days
Major adverse cardiovascular and cerebrovascular events (MACCE) event rate | Immediately after the procedure、30days、180days
Myocardial infarction rate | Immediately after the procedure、30days、180days
Rate of revascularization | Immediately after the procedure、30days、180days
Stent thrombosis rate | Immediately after the procedure、30days
Lumen diameter was obtained immediately after operation | Immediately after the procedure
Luminal area obtained immediately after operation | Immediately after the procedure